CLINICAL TRIAL: NCT05327491
Title: An Open-label, Randomized, Crossover Study in Healthy Volunteers to Compare the Pharmacokinetics of Sotorasib Administered as 1 or 2 Tablets
Brief Title: A Study in Healthy Volunteers to Compare the Pharmacokinetics of Sotorasib Administered as 1 or 2 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20210088
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-03

CONDITIONS: Healthy Participants
Keywords: Sotorasib; AMG 510
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence ABC (Experimental): Participants will be administered sotorasib orally in the following order:
  Period 1 - as 1 tablet (test 1) Period 2 - as 2 tablets (reference) Period 3 - as 1 tablet (test 2)
  Interventions: Drug: Sotorasib
- Treatment Sequence BAC (Experimental): Participants will be administered sotorasib orally in the following order:
  Period 1 - as 2 tablets (reference) Period 2 - as 1 tablet (test 1) Period 3 - as 1 tablet (test 2)
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Oral Tablet
  Other Names: AMG 510

SUMMARY:
The primary objective of the study is to compare the pharmacokinetics (PK) of sotorasib administered orally as 1 tablet under fasted conditions to sotorasib administered orally as 2 tablets under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants or female participants, between 18 and 60 years of age (inclusive), at the time of Screening.
* Body mass index, between 18 and 30 kg/m^2 (inclusive), at the time of Screening.
* Females of nonchildbearing potential.

Exclusion Criteria:

* Inability to swallow oral medication or history of malabsorption syndrome.
* History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Poor peripheral venous access.
* History or evidence, at Screening or Check in, of clinically significant disorder, condition, or disease, including history of myolysis, not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participants safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Labcorp Clinical Research Unit - Daytona Beach, Daytona Beach, Florida
  - Miami Research Associates LLC - Main Campus / Late Phase, South Miami, Florida
  - Labcorp Clinical Research Unit - Dallas, Dallas, Texas
  - Labcorp Clinical Research Unit - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 146 participants were enrolled with all participants randomized into Treatment Sequences AB and BA, including 14 participants that proceeded to receive Treatment C in the food effect substudy.
Groups:
- Treatment Sequence AB: Participants received a single oral dose of sotorasib under fasted conditions in the following order:
  Period 1 - as 1 tablet (test 1) on Day 1 Period 2 - as 2 tablets (reference) on Day 4
- Treatment Sequence BA: Participants received a single oral dose of sotorasib under fasted conditions in the following order:
  Period 1 - as 2 tablets (reference) on Day 1 Period 2 - as 1 tablet (test 1) on Day 4
- Treatment Sequence ABC: Participants who received treatment sequence AB in Periods 1 & 2 proceeded to receive a single oral dose of sotorasib administered as 1 tablet with a high-fat meal in Period 3 on Day 7.
- Treatment Sequence BAC: Participants who received treatment sequence BA in Periods 1 & 2 proceeded to receive a single oral dose of sotorasib administered as 1 tablet with a high-fat meal in Period 3 on Day 7.
Period: Periods 1 & 2
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Treatment Sequence ABC | Treatment Sequence BAC
Started | 73 | 73 | 0 | 0
Received at Least 1 Dose | 73 | 73 | 0 | 0
Completed | 72 | 72 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Miscellaneous | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 3 (Food Effect Substudy)
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Treatment Sequence ABC | Treatment Sequence BAC
Started | 0 | 0 | 7 | 7
Completed | 0 | 0 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Total
Number analyzed (Participants) | 73 | 73 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.6 (11.1) | 39.2 (10.74) | 38.4 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 67 | 59 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 29 | 59
  Not Hispanic or Latino | 43 | 44 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 41 | 44 | 85
  Black and African American | 27 | 25 | 52
  Asian | 3 | 4 | 7
  American Indian or Alaska Native | 1 | 0 | 1
  Multiple | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Period 1 and 2: Maximum Observed Plasma Concentration (Cmax) of Sotorasib
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on the 1st day of each period (Days 1 and 4)
Population: All participants who received at least 1 dose of sotorasib and had evaluable PK data and evaluable observations.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: All participants who received a single oral dose of sotorasib under fasted conditions as 1 tablet in either Period 1 or Period 2.
- Treatment B: All participants who received a single oral dose of sotorasib under fasted conditions as 2 tablets in either Period 1 or Period 2.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 145 | 145
ng/mL | 4170 (75.0) | 4340 (65.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — It was concluded that the test treatment is bioequivalent to the reference treatment if the 90% CI for the ratio of Geometric Least Squares Mean (GLSM) was completely contained within the predefined interval of (0.8000, 1.2500); Ratio of GLSM = 0.962, 90% CI 2-sided [0.880 to 1.053]

2. Primary Outcome: Period 1 and 2: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of Sotorasib
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of sotorasib and had evaluable PK data and evaluable observations.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 145 | 145
h*ng/mL | 15300 (56.2) | 15800 (54.6)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of GLSM = 0.968, 90% CI 2-sided [0.907 to 1.033]

3. Primary Outcome: Period 1 and 2: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of Sotorasib
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on on the 1st day of each period (Days 1 and 4)
Population: All participants who received at least 1 dose of sotorasib and had evaluable PK data and evaluable observations.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 144 | 145
h*ng/mL | 15500 (54.1) | 16100 (52.8)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of GLSM = 0.967, 90% CI 2-sided [0.908 to 1.029]

4. Secondary Outcome: Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an adverse event (AE) that started during or after dosing, or started prior to dosing and increased in severity after dosing within each period.
  Clinically significant laboratory tests, 12-lead electrocardiogram (ECG), or vital sign results as assessed by the Investigator were also recorded as adverse events.
Time Frame: Day 1 to Day 9
Measure: Count of Participants; unit: Participants
Groups:
- Treatment C: All participants who received a single oral dose of sotorasib as 1 tablet with a high-fat meal in Period 3.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 146 | 146 | 14
Participants | 3 | 10 | 0

5. Secondary Outcome: Period 3: Cmax of Sotorasib
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on the 1st day of Period 3 (Day 7)
Population: All participants who received at least 1 dose of sotorasib and had evaluable PK data and evaluable observations.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C
Number analyzed (Participants) | 14
ng/mL | 4530 (14.2)

6. Secondary Outcome: Period 3: AUClast of Sotorasib
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on on the 1st day of Period 3 (Day 7)
Population: All participants who received at least 1 dose of sotorasib and had evaluable PK data and evaluable observations.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment C
Number analyzed (Participants) | 14
h*ng/mL | 19000 (20.3)

7. Secondary Outcome: Period 3: AUCinf of Sotorasib
Time Frame: as for outcome 5
Population: All participants who received at least 1 dose of sotorasib and had evaluable PK data and evaluable observations.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment C
Number analyzed (Participants) | 14
h*ng/mL | 19100 (20.0)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 9
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/146 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/146 | 0/14
Other Adverse Events (participants affected / at risk) | 3/146 | 10/146 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=146) | Treatment B (N=146) | Treatment C (N=14)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT05327491/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05327491/SAP_001.pdf